CLINICAL TRIAL: NCT02032680
Title: Comparison of E-Health vs. In-Person Delivered Family Psychoeducation Treatment
Brief Title: Comparison of E-health vs. In-person Multi-Family Group (MFG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIR 13-332
Record Dates: First submitted 2013-12-30; First posted 2014-01-10 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophrenia and Related Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Web-based family psycho-education treatment (Experimental): The e-health/web-based intervention provides: three therapist facilitated group forums; a function to send facilitators questions; a library of previously answered questions; and a library of educational materials.
  Interventions: Behavioral: Web-based multi-family psychoeducational treatment
- In-persons Multi-Family Group Psycho-Education treatment (Active Comparator): This arm provides the evidence based multi-family psychoeducational treatment, termed Multi-Family Group Psycho-Education (MFG) that is the standard of care in the VA.
  Interventions: Behavioral: In-persons Multi-Family Group Psycho-Education treatment
- Treatment as Usual (Other): The Treatment as usual (TAU) group provides a benchmark against which to measure the impact of the two individual interventions (MFG & DSW) independent from each other. Through enhancements of TAU, such as regular monitoring which will be done in the assessment process and by the provision of information to VA psychiatrist when there are concerns or problems with the psychiatric status of their patients, we will be taking reasonable steps to ensure the safety of the participants who are assigned to TAU.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Web-based multi-family psychoeducational treatment — This intervention uses a website to provide multi-family psychoeducational treatment to Veterans and their family members or other supporters.
  Arms: Web-based family psycho-education treatment
Behavioral: In-persons Multi-Family Group Psycho-Education treatment — This intervention will provide the VA's evidence-based MFG. This intervention is delivered to Veterans and their families or other supporters using an in-person format.
  Arms: In-persons Multi-Family Group Psycho-Education treatment
Other: Treatment as usual (TAU) — Treatment as Usual (TAU) is considered the usual care at the VA. Participants assigned to be in the Treatment as Usual arm will complete assessments at all data collection time points, (baseline, 6, 12, and 15 months.) These participants will not receive any study treatment but will continue to receive their treatment as usual through the VA.
  Arms: Treatment as Usual

SUMMARY:
As specified in the VA Uniform Services Handbook, Family Psycho-Education (FPE) treatment must be available to all Veterans with schizophrenia who could benefit, and their family members. This includes those receiving care at Community Based Outpatient Clinics (CBOCs), and at Psychosocial Rehabilitation and Recovery Centers (PRRCs), whether provided on site, by referral, or by telemental health. However, less than 5% of VA medical centers offer FPE. Clearly, a major challenge is to devise ways to deliver mental health treatments and services to Veterans who need them in ways that meet their needs and preferences. The proposed project will compare the use of a website to deliver FPE to that of in-person delivered FPE. The findings could have profound implications for the VA's ability to improve the reach, use, appeal, and effectiveness of FPE for Veterans with schizophrenia, by using an e-health model that facilitates family involvement.

DETAILED DESCRIPTION:
In the VA Family Psycho-Educational (FPE) is a component of the Uniform Services standard for care of Veterans with schizophrenia and their family members. FPE includes single family variants, e.g., Behavioral Family Therapy, which is provided to individual families (consumer and family members); and multi-family variants, e.g., Multi-Family Group Psycho-Education (MFG-stands for 'Multi-Family Group Psycho-Education'), which is provided to multiple families (consumers and family members together) in a single treatment group. To promote the availability of FPE to all Veterans who could benefit, the VA began national trainings of clinicians in FPE. Despite this training, the proven effectiveness of FPE, and that it is the standard for care, it is not widely available to Veterans, is underutilized even where available, and can incur relatively high resistance from Veterans and families. Less than 5% of VA Medical Centers provide FPE. Further, even where it is available, it reaches a relatively small proportion of Veterans who could benefit. Barriers to receiving this treatment include the lack of appropriately trained clinicians, the need for Veterans and family members to travel to receive these services--this maybe a particularly important hurdle for a treatment that meets bi-weekly for a minimum of nine months--the tendency to avoid in-person treatment due to the stigma associated with seeking mental health treatment, and the difficulty of providing treatments after hours or on weekends when families are more likely be able to attend. It is important for the VA to have treatment delivery models that maximize the likelihood that all Veterans in need will receive interventions such as FPE, including Veterans residing in rural settings, and Veterans who avoid VA settings due to stigma. E-health delivery of services has been a focus of the VA as a way to overcome these barriers. Specialized web-based approaches have been studied and found to be successful for people with schizophrenia, and their families, and can deliver content that is intensive and engaging with reduced requirements for staff time.

The investigators' previous work has developed a model and guidelines to design e-health applications for persons with schizophrenia and others with cognitive impairments (e.g., Rotondi, VA Rehabilitation Research and Development D61804R), and developed a highly scalable intervention termed Schizophrenia On-line Access to Resources (SOAR) (Rotondi, R01 MH63484). SOAR incorporated FPE into a modernized model that: incorporates web-based delivery; provides the ability of users to individualize commitment and services to meet varied preferences and needs, in order to address prominent reasons for resistance to FPE; and is accessible from homes and smart phones. SOAR was highly successful at reducing illness symptoms for persons with schizophrenia and improving their and their family members' knowledge of the illness. The Daily Support Website (DSW) was created as the next iteration of SOAR, with improvements based on what was learned from the original trial.

The aims of this study are to conduct: 1) a non-inferiority randomized trial of the Daily Support Website (DSW) vs. in-person MFG vs. Treatment as usual (TAU) that compares the achievement of a personal goal, changes in severity of positive and negative psychiatric symptoms, and family psychological burden, during treatment and 3-months post-treatment 2) exploratory secondary analyses to identify Veteran and family characteristics that are associated with achievement of a personal goal, decreased levels of psychiatric symptoms and caregiver burden; 3) exploratory qualitative analyses to inform a larger implementation of the DSW by identifying barriers, facilitators, VA system requirements, etc. from clinicians providing the treatments, their supervisors, and participants. If successful, the DSW could substantially increase the options, availability, utilization, appeal, and effectiveness of FPE for Veterans and their families, thereby improving Veteran well-being, recovery, and Veteran and family quality of life.

ELIGIBILITY:
Inclusion Criteria:

Veterans will be included who:

* have a DSM-V (Diagnostic and Statistical Manual of Mental Disorders V) diagnosis of schizophrenia or schizoaffective disorder;
* are 18-75 years old; are not in another family treatment,
* and; are able to speak and read English at the 5th grade level.
* The primary support person for the Veteran must be 18 years old
* and able to speak and read English at the 5th grade level.

Exclusion Criteria:

* Unable to speak English
* or use necessary technology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armando J. Rotondi, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in all articles, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 month after publication.
Access Criteria: Outside investigators will follow VA procedures for approval and access.

REFERENCES:
- [Result] Rotondi AJ, Eack SM, Hanusa BH, Spring MB, Haas GL. Critical design elements of e-health applications for users with severe mental illness: singular focus, simple architecture, prominent contents, explicit navigation, and inclusive hyperlinks. Schizophr Bull. 2015 Mar;41(2):440-8. doi: 10.1093/schbul/sbt194. Epub 2013 Dec 27. PMID 24375458
- [Result] Rotondi AJ, Spring MR, Hanusa BH, Eack SM, Haas GL. Designing eHealth Applications to Reduce Cognitive Effort for Persons With Severe Mental Illness: Page Complexity, Navigation Simplicity, and Comprehensibility. JMIR Hum Factors. 2017 Jan 5;4(1):e1. doi: 10.2196/humanfactors.6221. PMID 28057610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 96 veterans screened, 78 met eligibility criteria.
Pre-assignment Details: Of the 78 who were screened and met eligibility criteria, 40 consented to participate in the study. 10 of the 40 dropped out before being assigned to an intervention arm. 30 were assigned to an intervention arm.
Groups:
- In-persons Multi-family Psycho-educational Treatment: This arm provides the evidence based multi-family psychoeducational treatment, termed Multi-Family Group (MFG) that is the standard of care in the VA.
  In-persons multi-family psycho-educational treatment: This intervention will provide the VA's evidence-based, in-person delivered, multi-family psychoeducational treatment, termed Multi-Family group (MFG). This intervention is delivered to Veterans and their families or other supporters using an in-person format.
Period: Overall Study
Arm/Group | Web-based Family Psycho-education Treatment | In-persons Multi-family Psycho-educational Treatment
Started | 22 | 8
Completed | 16 | 7
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Population: No TAU participants were recruited.
Groups:
- Web-based Family Psycho-education Treatment: The e-health/web-based intervention provides: three therapist facilitated on-line group forums; a function to send facilitators questions; a library of previously answered questions; and a library of educational materials.
  Web-based multi-family psychoeducational treatment: This intervention uses a website to provide multi-family psychoeducational treatment to Veterans and their family members or other supporters.
- Total: Total of all reporting groups
Arm/Group | Web-based Family Psycho-education Treatment | In-persons Multi-family Psycho-educational Treatment | Total
Number analyzed (Participants) | 22 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (10.9) | 51.4 (11.8) | 56.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 15 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 1 | 11
  White | 12 | 6 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 8 | 30
Participant Goal Attainment Scale [Mean (Standard Deviation); unit: units on a scale] — The scale ranges from 0 (worst) to 4 (best) and that by definition, at the time the goal was developed, each participant was at the base level, which was given a value of zero (0). At baseline, each participant in the DSW and MFG arms developed a goal that he or she would work on to achieve as part of their involvement in the study.
  units on a scale | 0 (0) | 0 (0) | 0 (0)

OUTCOME MEASURES:

1. Primary Outcome: Goal Attainment Scale
Description: At baseline, each participant developed a goal that she or he would work on to achieve as part of involvement in the study. Indicators of the 5 levels (0-4) of achievement, on the Goal Attainment Scale, were developed for each individual participant's goal, with each individual participant. The minimum was 0 (zero), the maximum was 4, and higher scores were better.
Time Frame: Outcome is assessed at 3, 6, and 12 months
Population: The analyses assessed the highest level that participants achieved on their goal, using the 5 point scale 0, 1, 2, 3, 4, with 4 being the highest achievement level The reported outcomes data indicates the highest level that a participant achieved on their goal during the study, regardless of which timepoint (3, 6, or 12 months) that this occurred.
Measure: Number; unit: percentage of participats
Arm/Group | Web-based Family Psycho-education Treatment | In-persons Multi-family Psycho-educational Treatment
Number analyzed (Participants) | 16 | 7
percentage of participats
  Highest level achieved was 1 | 6.25 | 14.29
  Highest level achieved was 2 | 37.5 | 0
  Highest level achieved was 3 | 18.75 | 28.57
  Highest level achieved was 4 | 37.5 | 57.14
Statistical Analysis 1: Comparison: Web-based Family Psycho-education Treatment vs In-persons Multi-family Psycho-educational Treatment; The two treatments were compared to see whether participants in one achieved a higher level on their goals (i.e., the maximum level achieved on the goal); Test type: Superiority; p = 0.3749, Cochran-Armitage Trend Test

ADVERSE EVENTS:
Time Frame: 15 months: from baseline (time 0) until the end of the intervention period (1 year), and then through a 3 month follow-up.
Arm/Group | Web-based Family Psycho-education Treatment | In-persons Multi-family Psycho-educational Treatment
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/8
Other Adverse Events (participants affected / at risk) | 0/22 | 0/8

LIMITATIONS AND CAVEATS:
The sample for each arm was relatively small. This was basically a pilot evaluation. A larger trial would be necessary to provide a full evaluation of each intervention and the relative advantages and disadvantages of each intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT02032680/Prot_SAP_000.pdf